CLINICAL TRIAL: NCT06193447
Title: Postoperative Early Mobilization and Affecting Factors in Patients Undergoing Open Heart Surgery: A Descriptive-Cross Sectional Study
Brief Title: Early Mobilization in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: Cardiac surgery
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Nursing Caries; Ambulation Difficulty
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None intervention — None intervention

SUMMARY:
This study was planned to determine the mobilization process and factors affecting this process in patients who underwent open heart surgery and were admitted to the cardiovascular surgery intensive care unit.

DETAILED DESCRIPTION:
Mobilization; It is defined as "standing up, walking, being able to move and walking around, especially after the operation, when the patient stands up and walks around". Postoperative mobilization is a basic human need and one of the basic principles of nursing care. In the postoperative period, with the delay of mobilization, the patient's insulin resistance increases, muscle weakness and muscle mass loss occur, problems in pulmonary functions are experienced and the risk of thromboembolism increases.

Surgery of patients admitted to cardiovascular ICUs after open heart surgery close monitoring afterwards, maintenance of cardio-respiratory functions, healing is supported. During care in the intensive care unit Preparation of materials that may be needed by the patient, general condition of the patient and vital information monitoring symptoms, performing breathing exercises, evaluating pain and management, monitoring fluid-electrolyte balance, monitoring hemodynamic parameters, surgical wound dressing, getting the patient up as soon as possible and in bed increasing mobility. In this process, while the mobilization process of the patients is planned, the patient's The general condition and tolerance regarding mobilization should be evaluated. patient's general Depending on the suitability of the condition, turning in bed, foot-leg exercises, deep breathing and gradual mobilization, such as cough exercises, sitting in bed, standing up, and walking inform the patient and the patient's family about the methods, plan the mobilization process, The patient should be evaluated before, during and after mobilization. Early postoperative mobilization is an important component of nursing care.

Early mobilization of patients after open heart surgery, although the recommendations to increase the mobility are getting stronger, the mobilization levels of the patients are still not at the desired level. Although studies examining the early mobilization process of patients after open heart surgery have been conducted so far, findings regarding the clinical factors affecting this process are very limited.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Staying in the cardiovascular intensive care unit for 24 hours or more

Exclusion Criteria:

* Being diagnosed with a psychiatric disorder
* Do not have active bleeding
* Do not have arrhythmia
* Reporting pain intensity of 4 or above on the Visual Analog Scale

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergoing open heart surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative mobilization level | Postoperative day 2
  Assessed with Intensive Care Units-Mobility Scale. The scale used to evaluate patient mobiility level on postoperative days. It consisted of 11 items with scoring, classification and explanation from 0 (zero) to 10 (ten), ranging from lying in bed/passive exercises to independent ambulation.
Pulse rate changes between before and after mobility | Twice: Before mobilization and after mobilization (5 minutes later)
  Assessed with a form which is created by authors. The form is containing the outcome both of before and after mobilization. These are calculated both time point.
Blood pressure (both of systolic and diastolic blood pressure) changes between before and after mobility | Twice: Before mobilization and after mobilization (5 minutes later)
  Assessed with a form which is created by authors. The form is containing the outcome both of before and after mobilization. These are calculated both time point.
Oxygen saturation changes between before and after mobility | Twice: Before mobilization and after mobilization (5 minutes later)
  Assessed with a form which is created by authors. The form is containing the outcome both of before and after mobilization. These are calculated both time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Ezgi Arslan, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all-authors within 1 month of receiving the request.